# GEOSCAN AND REMOTE GEO SMOKING STUDY: NEURAL AND BEHAVIORAL CORRELATES OF SMOKERS' EXPOSURE TO RETAIL ENVIRONMENTS

Principal Investigator Emily Falk, Ph.D.

Annenberg School for Communication

University of Pennsylvania

3620 Walnut Street, Philadelphia, PA 19104

215-573-9901

emily.falk@asc.upenn.edu

**Date** 09/20/2023

Funding Sponsor National Cancer Institute (NCI)

National Institutes of Health (NIH)

9609 Medical Center Dr, Rockville, MD 20850

800-422-6237

Protocol Number ClinicalTrials.gov Identifier: NCT04279483

IRB 850796

IRB Number ACC Identifier: UPCC# 08022

NIH Grant Number 1R01CA229305-01A1

# Screen B

#### Welcome to the Geo Smoking Study!

Thank you for your interest in the Geo Smoking Study at the University of Pennsylvania!

If you are taking this survey, you have already completed the first part of our screening process and have spoken with a study staff member about this task. We expect this survey to take about 30 minutes. First, you will be asked to read over the survey consent form. If you consent to completing the screening, you will be asked for information like your mailing address and your COVID-19 vaccination status. You will then be guided through the submission of your Google Timeline location history. We strongly recommend that you complete this survey on a laptop or desktop computer, as it will require you to switch tabs at different points.

## **Screening B Consent Form**

Primary Contact: Study Team

Phone:267-225-0399

Email: geo@falklab.org

**Emergency Contact: Alexandra Paul** 

Phone: 267-225-2341

Email: alexandra.paul@asc.upenn.edu

Principal Investigator: Dr. Emily Falk

Address: 3620 Walnut Street, Philadelphia, PA 19104

Phone: 215-573-9901

Fax: 215-898-2024

Email: emily.falk@asc.upenn.edu

The purpose of this screening task is to confirm your eligibility to participate in the Geo Smoking Study. Here, you will make an informed decision about whether you would like to complete the screening task.

#### What will I be asked to do?

This survey will guide you through the process of identifying the Google account associated with Google Maps on your phone, downloading a copy of your location history data, and sending it to the study team. You will also be asked to upload a photo of your COVID-19 vaccination card and provide your preferred shipping address.

#### What will you do with my information?

The information that you submit in this survey (name, address, date of birth, COVID-19 vaccination history, and mobile location history) will only be used by research staff in our laboratory for study purposes.

The study team will use your geolocation data to confirm that you live in the study area (anywhere in the states of PA, NJ, or DE), which is required for you to be eligible to participate in this study.

The team will look at the picture of your COVID-19 vaccination card to confirm that you meet the most up-to-date requirements to be considered fully vaccinated.

#### What will happen if I'm eligible for the study?

If the geolocation data and vaccination card that you submit in this screening confirm that you are eligible to enroll in the study, you will be mailed package containing study materials to the shipping address listed on this survey.

You will be given instructions for how to enroll in the full study and begin participating with the first online session once your study materials arrive. You can be paid up to \$95 once you complete the first online session, which includes payment for the first online session and all other tasks that were completed before the first online session (Intake call and Screening B). In other words, as long as the results of Screening Survey B confirm that you are eligible to participate, you will be paid for the screening and for the first online session after you complete the first online session. Total compensation for completing all stages of the full study is \$500.

If you decide not to participate in the full study, you may contact the study team at geo@falklab.org or by phone at 267-225-0399 to request that we delete the geolocation data file that you submitted. If we have not heard from you and you have not enrolled in the main study within 1 month of receiving the study materials, we will assume that you are no longer interested in participating and delete the geolocation data file that you submitted.

### What will happen if I'm not eligible for the study?

If you are found to be ineligible to participate in the main study, you will be contacted by the study team via email to inform you of this and provide you with instructions for turning off Google Timeline and uninstalling Google Maps. The study team will then delete the geolocation data file that you submitted.

#### **Potential Risks and Benefits**

Risks: There is always a risk of an unintentional breach of confidentiality about your information provided in the surveys or through the location tracking app, but we will make every effort to prevent this from happening. Your name and other identifiable information will be removed from all information we collect and will be replaced with a unique identification code. Additionally, we want you to be aware that this research is covered by a Certificate of Confidentiality from the National Institutes of Health. This means that the researchers cannot release or use information, documents, or samples that may identify you in any action or suit unless you say it is okay. Authorities also cannot provide any information, documents, or samples from this study as evidence unless you have agreed. This protection includes federal, state, or local civil, criminal, administrative, legislative, or other proceedings. An example would be that we would NOT provide your information in response to a court subpoena.

Potential benefits: There is no direct benefit to you for completing this screening task other than finding out if you are eligible to participate and potential compensation. We hope that the information learned from this study may benefit other people and further science by helping us to better understand the relationship between the brain, behavior, and exposure to daily environments.

#### Contacts

For any study-related questions or concerns, you may contact the study team (by email: geo@falklab.org or phone: 267-225-0399). The principal investigator for this study is Dr. Emily Falk, Ph.D. (emily.falk@asc.upenn.edu.

215-573-9901). You may also contact the Office of Regulatory Affairs with any questions, concerns or complaints at the University of Pennsylvania by calling (215) 898-2614.

Participation in this screening task is completely voluntary and if you decide not to complete it or want to stop at any point, there will be no penalty or loss of benefits to which you are otherwise entitled. If you do not want to complete the task, you can simply close your browser window now.

| Please note: You must be of the age of 21 or older to p | roceed |
|---------------------------------------------------------|--------|
|---------------------------------------------------------|--------|

| Please indicate whether you consent to complete the | <ul> <li>Yes, I wish to complete the online eligibility</li> </ul> |
|---|---|
| screening task in this survey: | screening survey for this research study. I have |
| · | read and understood the information above. |
| | No, I do not wish to complete the online |
| | eligibility screening survey for this research |
| | study. I will close my browser without answering |

any of the survey questions.

Sign here if you agree to complete this eligibility screening survey

#### OPTIONAL: Opt-out of the analysis of your Google Timeline data from before the study period

This component is only relevant if you are found to be eligible for the study. If you are found to be ineligible, all of your geolocation data will be deleted from our records regardless of your choice below.

If you have already installed and activated Google Timeline on your phone, we will have to download your location data from both before and during your participation in this study. By signing the previous consent form, you agree to the analysis of any Google Timeline data that we download. This data may include information on your location from both before and during the study period. However, you can prohibit analysis of your location data from before today, other than for the purpose of establishing study eligibility, without any consequences for your participation in the study. This means we would only use that information to determine if you live in the study area. If you opt out of allowing your past location data to be further analyzed, we will remove it from any future analyses and focus only on the data from the time between when you sign this form and when you finish participating.

To obtain a better understanding of your location patterns as they relate to your exposure to certain retail outlets, our research may benefit from analyzing all available data that might have been collected on your phone through Google Timeline.

However, if you wish, you can prohibit the study team from analyzing your location data from before the study period (i.e., before today), except for the purpose of establishing eligibility to participate in the study. Your decision in this matter does not impact or invalidate any other elements of the consent you provided above or the reimbursement you might receive for this research study. Please be aware that, regardless of your choice, your location data will be protected by a Certificate of Confidentiality from the National Institutes of Health. This means that no authority will have a legal means of accessing your location data or any other personally sensitive data without your permission.

If you wish to prohibit us from analyzing your data from before today, other than for the purpose of establishing eligibility, please copy or write the following sentence in the space below. Otherwise, leave the text box blank.

"Do not analyze my Google Timeline data from before the study period."